CLINICAL TRIAL: NCT02238808
Title: PRe-operative ESTradiOl Window of Opportunity Study in Post-Menopausal Women With Newly Diagnosed ER Positive Breast Cancer
Brief Title: A Study to See Whether Estrogen Can Slow the Growth of Some ER Positive Breast Cancers
Acronym: PRESTO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EER001
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Estrogen Receptor Positive Breast Cancer
Keywords: ER+ breast cancer; Luminal A; Estradiol
MeSH Terms: interventions — Estradiol; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estradiol treatment (Experimental): Estradiol 6 mg daily for 7-14 days
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Eligible participants will take 2 mg Estradiol 3 times daily for 7-14 days pre-surgery.
  Other Names: estrogen

SUMMARY:
Some breast cancers have estrogen receptors (ER+). The investigators know that some ER+ tumours can be cured by hormone therapy alone while other ER+ breast cancers cannot. Currently, there is no perfect way to tell these groups apart nor do the investigators know why some respond when others do not.

Research findings suggest that the two types of ER+ breast cancers differ in their response to estrogen with estrogen being toxic to one type and not the other. For those tumours that find estrogen toxic, this may explain why tumours only start to grow when estrogen levels decrease after menopause.

The purpose of this study is to see whether a two-week treatment of estrogen equal to pre-menopausal estrogen levels will decrease the rate at which patients' ER+ tumours grow. This will be done by comparing the growth rate in the tissue removed during standard of care surgery after patients have been treated with 7-14 days of estrogen prior to that surgery.

DETAILED DESCRIPTION:
Breast cancer is a heterogeneous disease that includes two ER+ genetic subtypes (luminal A and luminal B) that differ in their response to treatment.

Results from the Women's Health Initiative Trial showed that estrogen treated hysterectomized women with no prior history of breast cancer had a significant and persistent decrease in breast cancer incidence when compared to placebo treated participants. This implies that some ER+ breast cancers are in fact growth inhibited by estrogens and are not growth promoted.

The hypothesis of this study is that some ER+ breast cancers (luminal A) are actually sensitive (growth inhibited) by estrogen.

Objectives:

1. To assess changes in breast cancer proliferation after a 7-14 day trial of estradiol in newly diagnosed estrogen receptor positive post-menopausal breast cancer patients prior to surgery.
2. Exploratory analysis of biologic correlates with comparison to available genotyping tests.

This is an open-label single group assignment pilot study for safety/efficacy and exploratory biologic correlates

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Estrogen receptor positive (ER+) breast cancer
* HER2 negative breast cancer
* Post-menopausal by greater than 5 years
* No previous hormonal replacement therapy
* Low to intermediate histologic grade
* ECOG Performance status of 0 of 1
* Adequate hematological, renal and hepatic function is required
* Ability to take oral medication
* Patient must have adequate tissue for diagnosis, biomarkers and Ki67 assays

Exclusion Criteria:

* Pre-menopausal women
* Locally advanced or metastatic breast cancer
* Current, previous or planning for pre-operative treatment with chemotherapy, hormone therapy including corticosteroids, radiation therapy for malignancy or other condition
* Known hypersensitivity or intolerance to estradiol
* Ischemic changes on baseline electrocardiogram
* Symptomatic but untreated cholelithiasis
* History of deep vein thrombosis, pulmonary embolism, stroke, acute myocardial infarction, congestive cardiac failure, untreated hypertension or known inherited hypercoagulable disorder
* Undiagnosed abnormal vaginal bleeding or prior history of endometrial cancer
* Untreated metabolic disturbances (glucose > 15.0 mmol/L and triglycerides > 400 mg/dL)
* Current treatment with drugs known to be moderate or strong inhibitors of inducers of isoenzyme CYP3A4
* The time between study enrolment and definitive breast surgery is not sufficient for administration of at least 7 days of estradiol

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07-30 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To assess changes in breast cancer proliferation after a 7-14 day trial of estradiol in newly diagnosed estrogen receptor positive post-menopausal breast cancer patients prior to surgery. | end of 7-14 day treatment with estradiol

SECONDARY OUTCOMES:
Exploratory analysis of biologic correlates with comparison to available genotyping tests | end of 7-14 day treatment with estradiol
Analysis of recurrence/survival data based on initial Ki67 response to 7-14 day trial of estradiol. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hugh, MD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No